CLINICAL TRIAL: NCT05560373
Title: The Effect of Huperzine A Injection on Postoperative Cognitive Dysfunction in Patients With Aneurysmal Subarachnoid Hemorrhage: a Pilot Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wanbangde Pharmaceutical Group Co., LTD (Industry)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220784
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Cognitive Dysfunction in Patients With Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: interventions — huperzine A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The operation group-The treatment group (Experimental): after operational treatment: ①the best basic treatment ②i.m. huperzine A injection (0.2mg), qd, 8d.
  Interventions: Drug: Huperzine A injection, operational treatment, the best basic treatment
- The operation group-The control group (Other): after operational treatment: ①the best basic treatment
  Interventions: Other: operational treatment, the best basic treatment
- The intervention group-The treatment group (Experimental): after interventional treatment: ①the best basic treatment ②i.m. huperzine A injection (0.2mg), qd, 8d.
  Interventions: Drug: Huperzine A injection, interventional treatment, the best basic treatment
- The intervention group-The control group (Other): after interventional treatment: ①the best basic treatment
  Interventions: Other: Interventional treatment, the best basic treatment

INTERVENTIONS:
Drug: Huperzine A injection, operational treatment, the best basic treatment — intramuscular
  Arms: The operation group-The treatment group
Other: operational treatment, the best basic treatment — other
  Arms: The operation group-The control group
Drug: Huperzine A injection, interventional treatment, the best basic treatment — intramuscular
  Arms: The intervention group-The treatment group
Other: Interventional treatment, the best basic treatment — other
  Arms: The intervention group-The control group

SUMMARY:
Under the premise of basic treatment, to explore the improvement effect of huperzine A injection on short-term and long-term neurocognitive dysfunction in patients with aneurysmal subarachnoid hemorrhage after interventional/surgical treatment.

DETAILED DESCRIPTION:
Description: This is a randomized, controlled, single center, exploratory clinical trial. The subjects are divided into surgical treatment group and interventional treatment group. Each group is divided into test group and control group. The test group is given huperzine A injection (0.2mg/dose) every day, intramuscular injection, for a total of 8 days, and basic treatment is given at the same time; The control group was given basic treatment, and did not receive other neurotrophic drugs except basic drugs. This clinical trial is to evaluate the effect of huperzine A injection on the improvement of postoperative cognitive dysfunction in patients with aneurysmal subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70;

  * The patients were proved to be aneurysmal subarachnoid hemorrhage by imaging examination (head CT, CT angiography (CTA), whole brain angiography (DSA));

    * Hunt Hess was graded I-III at admission;

      * The patients were treated with endovascular therapy or craniotomy and clipping surgery;

        * The time from the onset of aSAH symptoms to admission ≤ 72 hours; ⑥ The subject himself or the guardian of the subject knew and voluntarily signed the informed consent form.

Exclusion Criteria:

* Non aneurysmal subarachnoid hemorrhage;

  * Cognitive dysfunction existed before onset;

    * Patients with angina pectoris, bronchial asthma, mechanical intestinal obstruction, liver and kidney insufficiency, and urinary tract obstruction;

      * Complicated with other nervous system diseases, including nervous system degenerative diseases (Alzheimer's disease, Parkinson's disease, Lewy body dementia, frontotemporal dementia, etc.), neuromyelitis optica, epilepsy, central nervous system infection (such as AIDS, syphilis, etc.), brain traumatic dementia, etc;

        * Psychotic patients, according to DSM-IV-TR standards, including schizophrenia or other mental diseases, bipolar disorder, major depression or delirium;

          * Other cholinesterase inhibitor drugs are being used; ⑦ There are uncorrectable visual and auditory disorders, and neuropsychological tests and scales cannot be completed;

            * Have unstable or serious heart, lung, liver, kidney and hematopoietic system diseases;

              * Pregnant or lactating women and women of childbearing age without reliable contraception, and there is no evidence of negative pregnancy; ⑩ Patients who cannot be followed up as required during the study period; ⑪ Those who are allergic to the test drug; ⑫ Those who have participated in other clinical trials in recent 3 months; ⑬ Patients who are not suitable to participate in the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Mini Mental Status Examination（MMSE ） | 90 days after discharge
  The seven items in the scale were used for scoring, and the degree of intellectual status and cognitive impairment before treatment, during follow-up and after treatment were compared within and between groups. The higher the score, the better the intellectual state of the subjects.

SECONDARY OUTCOMES:
Hospital anxiety and depression Scale（HADS） | Screening period (day -4 to day 0), day 8, 30 days after discharge, 90 days after discharge and 180 days after discharge
  The anxiety and depression subscales of the Hospital Anxiety and Depression Scale were used to screen the anxiety and depression of the subjects before treatment, at the end of medication and at the visit period after discharge, and the intra group and inter group comparisons were made. The higher the score, the more serious the anxiety or depression.
The Short Form-36 Health Survey | Screening period (day -4 to day 0), 30 days after discharge, 90 days after discharge and 180 days after discharge
  Calculate the eight items in the scale. Before and after treatment, the scores of each items and the total score of body and psychology were compared within and between groups.
Modified Rankin Score | Screening period (day -4 to day 0), day 8, 30 days after discharge, 90 days after discharge and 180 days after discharge
  The functional recovery outcomes before treatment, at the end of medication and at the visit period after discharge were evaluated by using the modified Rankin scale, and compared within and between groups. The higher the score, the worse the functional recovery.
Biological sample detection | Screening period (day -4 to day 0), day 2, day 3, day 8
  Biological samples were tested during the screening period, during the medication period, and after the medication period to obtain drug metabolomics analysis data and disease biomarker data, and intra-group and inter-group comparisons were performed.
Mini Mental Status Examination（MMSE ） | Screening period (day -4 to day 0), day2, day 3, day 8, 30 days after discharge and 180 days after discharge
  The seven items in the scale were used for scoring, and the degree of intellectual status and cognitive impairment before treatment, during follow-up and after treatment were compared within and between groups. The higher the score, the better the intellectual state of the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No